CLINICAL TRIAL: NCT04037345
Title: A Open, Single-center, Phase 1 Trial to Evaluate Safety and Explore Efficacy of SMUP-IA-01 in Patients With Knee Osteoarthritis
Brief Title: Evaluate Safety and Explore Efficacy of SMUP-IA-01 in Patients With Knee Osteoarthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medipost Co Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MP-SMUP-IA-01-P01
Record Dates: First submitted 2019-07-17; First posted 2019-07-30 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2020-08

CONDITIONS: Knee Osteoarthritis
Keywords: human umbilical cord blood derived mesenchymal stem cells; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SMUP-IA-01(low-dose) (Experimental): A single knee administration of SMUP-IA-01 (low-dose, 4.0 x 10^6 cells/2mL) (2 ml of 1% sodium hyaluronate injection is administered before administration of SMUP-IA-01)
  Interventions: Biological: SMUP-IA-01(low-dose)
- SMUP-IA-01(mid-dose) (Experimental): A single knee administration of SMUP-IA-01 (mid-dose, 1.0 x 10^7 cells/2mL) ( 2 ml of 1% sodium hyaluronate injection is administered before administration of SMUP-IA-01)
  Interventions: Biological: SMUP-IA-01(mid-dose)
- SMUP-IA-01(high-dose) (Experimental): A single knee administration of SMUP-IA-01 (high-dose, 2.0 x 10^7 cells/2mL) (2 ml of 1% sodium hyaluronate injection is administered before administration of SMUP-IA-01)
  Interventions: Biological: SMUP-IA-01(high-dose)

INTERVENTIONS:
Biological: SMUP-IA-01(low-dose) — A single knee administration of SMUP-IA-01(low-dose, 4.0 x 10^6 cells/2mL)
  Other Names: Human umbilical cord blood-derived mesenchymal stem cells
  Arms: SMUP-IA-01(low-dose)
Biological: SMUP-IA-01(mid-dose) — A single knee administration of SMUP-IA-01(mid-dose, 1.0 x 10^7 cells/2mL)
  Other Names: Human umbilical cord blood-derived mesenchymal stem cells
  Arms: SMUP-IA-01(mid-dose)
Biological: SMUP-IA-01(high-dose) — A single knee administration of SMUP-IA-01(high-dose, 2.0 x 10^7 cells/2mL)
  Other Names: Human umbilical cord blood-derived mesenchymal stem cells
  Arms: SMUP-IA-01(high-dose)

SUMMARY:
This clinical trial is performed with patients with knee osteoarthritis who were radiologically diagnosed with Kellgren-Lawrence (K&L) grade 2 or 3. Subjects who voluntarily signed consent form and met inclusion/exclusion criteria, were evaluated eligible and participated in this trial. Investigator selected knee to be evaluated (right or left) and administered investigational product to selected knee on Day 1.

A total of 3 or 6 subjects will be enrolled in low-dose or mid-dose group each, and 6 subjects will be enrolled in high-dose group. The study used a dose escalation scheme (from low-dose to high-dose) to determine the maximum tolerated dose (MTD).

DETAILED DESCRIPTION:
All subjects in each dose-group will visit 1 month* (visit 5, 1 month±5 days) after administration of investigational product to evaluate dose limit toxicity (DLT) and determine whether to drop or proceed to next dose level.

Total 5 visit (1week, 1 month, 2 months, 3 months, 6 months) until 6 months after administration of investigational product is planned to assess safety through vial sign, laboratory tests, and exploratory efficacy of IP will be assessed through Western Ontario and McMaster Universities osteoarthritis index (WOMAC), 100-mm visual analogue scale (VAS) and International Knee Documentation Committee (IKDC) subjective knee evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female over 19 years of age
2. Subject with knee osteoarthritis (OA) and were diagnosed K&L grade 2 or 3 in radioactive examination at time of screening
3. Subject with more than 40mm joint pain on the 100-mm VAS, at the time of screening
4. Subject who were diagnosed as knee osteoarthritis by American College of Rheumatology (ACR) guideline criteria, at the time of screening
5. Subject with Body mass index (BMI) ≤35 kg/m2 at the time of screening
6. Subject with ligament instability ≤Grade II (grade o: no ligament instability, grade I: 0 ~ 5㎜, grade Ⅱ: 5 ~ 10 ㎜, grade Ⅲ: > 10 ㎜) at the time of screening
7. Subject who agree to maintain contraception during study period
8. Subject who voluntarily agreed to participate in the study, and signed informed consent

Exclusion Criteria:

1. Subject with myocardial infarction, congestive heart failure, and other severe heart disease or hypertension (or medical history of hypertension) that are not controlled below 140/90mmHg even with treatment with more than three(3) antihypertensive drugs
2. Subject with serious medical conditions other than cardiovascular disease
3. Subject with, or with a medical history of auto-immune diseases
4. Subject with an infection that requires parenteral antibiotic administration.
5. Subject with a medical history of mental disorder or epilepsy
6. Subject with chronic inflammatory joint diseases such as rheumatoid arthritis (e.g., osteoarthritis with infectious joint disease, gouty arthritis, and osteoarthritis)
7. Subject who had surgery or radiation therapy on knee joint area, or have not recovered from side effects of knee joint surgery within 12 weeks before screening
8. Subject who are pregnant or lactating
9. Subject abuse alcohol 10 times a week or smoke 25 cigarettes a day
10. Subject who were diagnosed with cancer within 5 years before screening
11. Subject who particiapted in another clinical trial within 4 weeks before screening of this clinical trial
12. Subject who were administered with immunosuppressnats such as cyclosporin A or azathioprine within 6 weeks before screening
13. Subject who had intra-articular administration such as sodium hyaluronate injections within 6 month before screening
14. Subject who are suffering from skin disease or considered inappropriate for injection in the injection site
15. Subject who has history of allergic response to hyaluronate injections or DMSO (cryopreservative) or Gentamicin (antibiotics)
16. Subject who are consiered inappropriate for MRI assessment with Tesla higher than 3.0
17. Subject with medical history of cell therapy product administration or are scheduled to administer other cell therapy product
18. Subject who principal investigator (PI) considers inappropriate to participate in the study due to any reasons other than those listed above

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2020-11-12 (Actual)

PRIMARY OUTCOMES:
Change of total score in WOMAC (Western Ontario and McMaster University Osteoarthritis Index) compared to baseline at 6 months after treatment | Baseline, Month 6
  Change of total scorein WOMAC compared to baseline at 6 months after treatment. WOMAC consists of three subscales: pain, stiffness, and physical function, and is performed on baseline (visit 2) and final (Visit 8) visits. Total of 24 questions are evaluated with 5 questions for pain, 2 questions for stiffness, and 17 questions for physical function. Each question is scored between 0 point (no symptom) ~ 4 points (severe symptoms) scale, and the total score is between 0 point (no symptoms) ~ 96 points (higher score representing worse symptoms).

SECONDARY OUTCOMES:
Change of score in WOMAC three subscales (Pain, stiffness, physical function)compared to baseline at 6 months after treatment | Baseline, Month 6
  The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68).
Change of score in 100 mm VAS (Visual Analogue Scale) compared to baseline | Baseline, Month 1, Month 2, Month 3, Month 6
  The VAS is a horizontal line, 100 mm in length and anchored by word descriptors at each end (no pain, very severe pain). The patient marks on the line at the point that represents their current state. The VAS score is determined by measuring in millimeters from the left hand end to the point of the mark. The score ranges from "0" or no pain to "100" very severe pain.
Change of score in IKDC(International Knee Documentation Committee)compared to baseline | Baseline, Month 1, Month 2, Month 3, Month 6
  Change of score in IKDC compared to baseline. IKDC subjective knee evaluation consists of three categories: symptoms, sports activities, and functions. For each category, there are 7 questions for symptoms, 2 questions for sports activities, and 2 questions for functions, a total of 11 questions for evaluation. The scores for each category are summed up and divided into 87, which is the maximum score possible, and then is evaluated by converting it into a scale of 100 points. Higher score indicates better function and less symptoms for the knee.
Change of score in WORMS(Whole-Organ Magnetic Resonance iMaging Score) compared to baseline at 6 months after treatment | Baseline, Month 6
  For structural and tissue evaluation of knee, MRI image of detailed knee parts are graded from min. 0 to max. 6. Lower number indicate normal status
Change in K&L(Kellgren-Lawrence) grade compared to the baseline at 3 months and 6 months after treatment | Baseline, Month 3, Month 6
  The K & L grade is 0 to 4 Grade, which means that the higher the grade, the greater the joint damage and the stenosis of the joint.
Change in joint space width compared to the baseline at 3 months and 6 months after treatment | Baseline, Month 3, Month 6
  Evaluation of disease progression in target knee as ascertained by change from baseline in joint space width (JSW) determined using radiography
Change in mechanical axis, anatomical axis compared to the baseline at 3 months and 6 months after treatment | Baseline, Month 3, Month 6
  The degree of deformation of the lower half of the body is measured by measuring the angles of the mechanical axis and the anatomical axis with respect to the vertical axis. Mechanical axis: A line connecting the femoral head center point and the ankle joint center point. Anatomical axis: The middaphyseal line of the femur and tibia.

CONTACTS AND LOCATIONS:
Overall Officials: Myungchul Lee, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea